CLINICAL TRIAL: NCT04422301
Title: Correlation Between Heart Rate Variability and Performance in Eccentric Resistance Training Associated With Partial Blood Flow Restriction: a Randomized Clinical Trial
Brief Title: Correlation Between HRV and Performance in Eccentric Resistance Training Associated With Partial Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franciele Marques Vanderle (Other)
Responsible Party: Sponsor-Investigator, Franciele Marques Vanderle, Clinical Professor, Paulista University
Organization: Paulista University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Unesp
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Exercise
Keywords: resistance training; vascular occlusion; performance; autonomic nervous system; recovery of physiological function
MeSH Terms: conditions — Motor Activity | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High intensity eccentric training (Experimental): High intensity eccentric training high intensity (80% isometric peak) eccentric training of the knee extensors in the isokinetic will be performed during 6 weeks, 3 times a week.
  eccentric exercise with blood flow restriction High/low intensity eccentric training group (80% and 40% of isometric peak torque) with or not blood flow restriction.
  Interventions: Other: Blood flow restriction
- High intensity eccentric training with blood flow restriction (Experimental): High intensity eccentric training with blood flow restriction high intensity (80% isometric peak) eccentric training of the knee extensors in the isokinetic associated with a pressure cuff placed in the proximal thigh (40% of absolute occlusion pressure) will be performed during 6 weeks, 3 times a week. eccentric exercise with blood flow restriction High/low intensity eccentric training group (80% and 40% of isometric peak torque) with or not blood flow restriction
  Interventions: Other: Blood flow restriction
- Low intensity eccentric training (Experimental): A low intensity (40% isometric peak) eccentric training of the knee extensors in the isokinetic will be performed during 6 weeks, 3 times a week. eccentric exercise with blood flow restriction High/low intensity eccentric training group (80% and 40% of isometric peak torque) with or not blood flow restriction.
  Interventions: Other: Blood flow restriction
- Low intensity eccentric training with blood flow restriction (Experimental): A low intensity (40% isometric peak) eccentric training of the knee extensors in the isokinetic associated with a pressure cuff placed in the proximal thigh (40% of absolute occlusion pressure)will be performed during 6 weeks, 3 times a week. eccentric exercise with blood flow restriction High/low intensity eccentric training group (80% and 40% of isometric peak torque) with or not blood flow restriction.
  Interventions: Other: Blood flow restriction

INTERVENTIONS:
Other: Blood flow restriction — an alternative method to produce strength and muscle hypertrophy with lower intensities

SUMMARY:
Studies on resistance training (RT) associated with blood flow restriction (BFR) is an alternative method of gaining strength and hypertrophy muscle. However, there is a gap correlated to autonomic repercussion of BFR and performance. Thus, it becomes relevant to investigate this type of training in post-exercise. Objective: investigate and compare autonomic and performance responses of 6 weeks of eccentric RT with different intensities associated or not to BFR in healthy youngsters. Method: This is a randomized clinical trial including 60 healthy men aged 18-35 years, divided into four groups according to exercise intensity and BFR: 80% without BFR, 40% without BFR, 80% with BFR and 40% with BFR. Exercise intensity will be determined by the peak of excentric torque on the isokinetic dynamometry method and by the BFR, as being 40% of the intensity required for the complete examination of the blood flow evaluated by Doppler. Participants will do an eccentric femoral quadriceps muscle exercise session on the isokinetic dynamometer according to the previously randomized group. For recovery analyzes, it will be used: the root-mean-square of the successive normal sinus RR interval difference (rMSSD); high frequency (HF) ms²; HF(nu) and the standard deviation of instantaneous beat-to-beat interval variability (SD1). For performance, it will be used the single leg hop test.

For data analysis of the population profile, the descriptive statistical method will be used and the results will be presented with values of means, standard deviations, median and confidence interval. Initially, participants from all study groups will be dichotomized at each performance outcome (muscle strength test on the isokinetic dynamometer and vertical jump test) as "improvement" or "without improvement" in order to demonstrate the behavior of the responses obtained during the training, that is, whether the individual responded to the RT or not. It is worth mentioning that this qualitative analysis will be performed considering the data obtained from the initial, intermediate and final evaluation.

The dichotomization of the results of the functional tests will be performed by the typical error of the sample measurement for each test. It will be considered as "improvement" if the participant presents gains in tests above the typical error of the measure. The values obtained from the initial, intermediate and final evaluation will be analyzed independently.

Subsequently, the weekly average of the vagal indices (rMSSD, HF and SD1) will be performed in the baseline moment and after 6 weeks of RT moment of each study group. In the sequence, the performance parameters will be correlated with the autonomic parameters in the respective groups. Pearson or Spearman correlation test will be used according to the normality of the data. The level of significance will be p <0.05 for all tests. The statistical program SPSS (Statistical Package for the Social Sciences) will be used for the analyzes.

ELIGIBILITY:
Inclusion Criteria:

* male sex;
* healthy;
* aged between 18 and 35 years

Exclusion Criteria:

* smokers
* alcoholics;
* use drugs that influenced cardiac autonomic activity;
* cardiovascular, metabolic or endocrine diseases.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Performance | Baseline
  Single Leg Hop Test
Performance | up to 3 weeks
  Single Leg Hop Test
Performance | after 6 weeks from baseline.
  Single Leg Hop Test
HRV - rMSSD | during the 6 weeks of training
  rMSSD (square root of the mean squared differences of successive N-N intervals)
HRV - SD1 | during the 6 weeks of training
  SD1 - the standard deviation of instantaneous beat-to-beat interval variability
HRV - HF (ms²) | during the 6 weeks of training
  HF (ms²) - (high frequency)
HRV -HF (nu) | during the 6 weeks of training
  HF (nu) - (high frequency)

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil